CLINICAL TRIAL: NCT03083782
Title: A Phase I, Open-Label, Crossover, Drug Interaction Study of Apixaban With Cyclosporine and Tacrolimus in Healthy Volunteers
Brief Title: Drug Interaction Study of Apixaban With Cyclosporine and Tacrolimus
Acronym: ACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10570; BMS-CV185-567 (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2017-03-06; First posted 2017-03-20 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Venous Thromboembolism; Pharmacokinetics; Healthy
Keywords: Apixaban; Cyclosporine; Tacrolimus; Cytochrome P450 CYP3A4; Permeability Glycoprotein P-gp; Breast cancer resistance protein BCRP; Factor Xa Inhibitors; Anticoagulants; Enzyme Inhibitors
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Cyclosporine; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Intervention Model: Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment A: Apixaban alone (Active Comparator): Oral apixaban will be administered in healthy volunteers to define baseline apixaban pharmacokinetics
  Interventions: Drug: Apixaban alone
- Treatment B: Cyclosporine with apixaban (Experimental): Oral cyclosporine will be administered to steady state in healthy volunteers followed by a single oral dose of apixaban to define apixaban pharmacokinetics in the presence of cyclosporine
  Interventions: Drug: Cyclosporine; Drug: Apixaban
- Treatment C: Tacrolimus with apixaban (Experimental): Oral tacrolimus will be administered to steady state in healthy volunteers followed by a single oral dose of apixaban to define apixaban pharmacokinetics in the presence of tacrolimus
  Interventions: Drug: Tacrolimus; Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban alone — A single dose of 10 mg apixaban administered orally at 0H on Day 1.
  Other Names: ELIQUIS
  Arms: Treatment A: Apixaban alone
Drug: Cyclosporine — Once daily dose of 100 mg cyclosporine administered orally on Days 1 to 3.
  Other Names: NEORAL
  Arms: Treatment B: Cyclosporine with apixaban
Drug: Tacrolimus — Once daily dose of 5 mg tacrolimus administered orally on Days 1 to 3.
  Other Names: PROGRAF
  Arms: Treatment C: Tacrolimus with apixaban
Drug: Apixaban — A single dose of 10 mg apixaban administered orally on Day 3 immediately following cyclosporine
  Other Names: ELIQUIS
  Arms: Treatment B: Cyclosporine with apixaban
Drug: Apixaban — A single dose of 10 mg apixaban administered orally on Day 3 immediately following tacrolimus
  Other Names: ELIQUIS
  Arms: Treatment C: Tacrolimus with apixaban

SUMMARY:
This study aims to evaluate the pharmacokinetics (PK) of apixaban when co-administered with cyclosporine and tacrolimus in healthy volunteers. The study participants will receive apixaban alone, cyclosporine followed by apixaban and tacrolimus followed by apixaban.

DETAILED DESCRIPTION:
Life- and graft-threatening complications in solid organ transplant patients have been greatly reduced due to the potent immunosuppressive agents like calcineurin inhibitors (CNI) that include cyclosporine and tacrolimus. Venous thromboembolism (clots in legs or lungs) in transplant recipients is often difficult to manage due to polypharmacy and potential for drug interactions. More than 90% of renal transplant (RT) recipients are maintained on a CNI-based immunosuppressive regimen. Cyclosporine is an inhibitor of many metabolic pathways including cytochrome P450 (CYP) 3A4, permeability glycoprotein (P-gp) and, breast cancer resistance protein (BCRP). Tacrolimus shares some of the distributive and metabolic pathways of cyclosporine. Apixaban is a combined substrate of CYP3A4, P-gp and, BCRP and thus has the potential for drug interactions with cyclosporine and tacrolimus. Apixaban levels that are too high or too low could be a problem for transplant patients. The purpose of this study is to determine what happens to apixaban blood levels when given in combination with cyclosporine or tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy male or female between ages 18-55 (inclusive) at the screening visit
2. Have a body mass index (BMI) ≥ 19 and ≤ 33 (inclusive)
3. Be a female subject, subject

   1. Can be of childbearing potential and must demonstrate a urine β-hCG level consistent with the non-pregnancy state and agree to use an acceptable method of birth control throughout the study.
   2. Can be of non-childbearing potential.
4. Be a nonsmoker for at least approximately 6 months
5. Have serum creatinine level < 1.5 mg/dL
6. Have a prothrombin time (PT) and activated partial thromboplastin time (PTT) level below the upper limit of normal
7. Have platelet count within normal limits
8. Be willing to refrain from the use of anticoagulants and antiplatelet medications including aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) during the entire period of study participation
9. Be willing to comply with trial restrictions

Exclusion Criteria:

1. Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures), dermatologic or psychiatric abnormalities or diseases
2. Has history of cancer (excluding treated cutaneous squamous or basal cell carcinoma of >3 years previous)
3. Has history of venous or arterial thromboembolic disease
4. Has a history of a major bleeding event (defined as: (i) symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or (ii) a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells) within 6 months prior to screening visit
5. Has had major surgery within 6 months prior to screening visit
6. Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies for 2 weeks prior to trial start date until the post-trial visit
7. Is unable to refrain from using any drugs or substance known to be inhibitors or inducers of cytochrome P450 (CYP) enzymes including grapefruit products for 2 weeks prior to dosing and throughout the study, until the post-trial visit
8. Has a history of illicit drug abuse within six months prior to screening visit
9. Pregnant or lactating
10. Consumes greater than 3 glasses of alcoholic beverages per day and cannot refrain from alcohol for the duration of the trial
11. Has a history of significant multiple and/or severe allergies (e.g. food, drug), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
12. Has known anaphylactic or severe systemic reactions to any components of study drugs (including apixaban, cyclosporine or tacrolimus) or contraindication to the administration of study drugs
13. Has moderate or severe hepatic disease or other clinically relevant bleeding risk
14. Has positive history for hepatitis B surface antigen, hepatitis C or HIV
15. Use of any drugs or products which at the discretion of the investigator would increase bleeding risk
16. Is considered inappropriate for participation by the investigator for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Apixaban area under the plasma concentration curve between 0 and 72 hours (AUC(0-72)). | Days 1-4 (Treatment A), Days 3-6 (Treatment B & C)
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm.
Apixaban peak plasma concentration (Cmax) | Days 1-4 (Treatment A), Days 3-6 (Treatment B & C)
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm.

SECONDARY OUTCOMES:
Safety and tolerability of apixaban when co-administered with cyclosporine assessed by capturing adverse events and laboratory safety tests | Day 1-4 (Treatment A), Day 1-6 (Treatment B & C)
  Safety and tolerability of apixaban when co-administered with cyclosporine based on adverse events reports and the results of vital sign measurements, electrocardiogram, physical examinations, and clinical laboratory tests
Safety and tolerability of apixaban when co-administered with tacrolimus assessed by capturing adverse events and laboratory safety tests | Day 1-4 (Treatment A), Day 1-6 (Treatment B & C)
  Safety and tolerability of apixaban when co-administered with tacrolimus based on adverse events reports and the results of vital sign measurements, electrocardiogram, physical examinations, and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes